CLINICAL TRIAL: NCT00544245
Title: Is Monitoring Activity Important for Short- and Long-term Weight Loss?
Acronym: UHPAWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: The Apex Fitness Group (Unknown); Bookman Publishing Company (Unknown)
Responsible Party: Charles Alan Titchenal, PhD, Assistant Professor, Human Nutrition, Food & Animal Sciences Dept., University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 437846
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Overweight and Obesity
Keywords: overweight; obesity; accelerometer; pedometer; energy balance; weight loss; weight maintenance
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Self monitoring of estimated energy balance — Participant estimation of energy intake and energy expenditure

SUMMARY:
This study is comparing the effectiveness of two techniques for monitoring physical activity and energy balance on long-term weight management (two years). The focus is on weight loss, prevention of weight gain, and the maintenance of a healthy weight over time. It is expected that both techniques will benefit long-term weight management.

DETAILED DESCRIPTION:
The major objective of this study is to determine if two techniques for monitoring physical activity and energy balance promote the maintenance of weight loss in healthy overweight and obese individuals. The study compares two approaches designed to help individuals monitor physical activity and to adjust their calorie intake to maintain a reasonable energy balance (bodybugg® & Step Diet Book systems). Full subject participation in the study spans two years. Participants periodically report to a pre-arranged location to be measured by a qualified fitness professional for height, weight, circumferences, and estimated body fat using a bioelectric impedance scale (body fat scale).

ELIGIBILITY:
Inclusion Criteria:

* Desire to lose weight
* Height: 60-76 inches
* BMI 27-40
* Healthy

Exclusion Criteria:

* Currently enrolled in a weight loss program
* Currently under medical care for obesity treatment
* Using drug, supplement, or similar treatment to promote weight loss
* Have undergone bariatric surgery or have breast implants
* Intend to have surgery within the next 24 months
* Have had an eating disorder
* Are pregnant, breast-feeding, or plan to become pregnant within 24 months
* Are planning an extended vacation, absence, or relocation within 24 months
* Use tobacco products
* Frequently consume 2 or more alcoholic drinks per day
* Use illegal drugs, steroids, or growth hormone
* Use any appetite-affecting medications
* Are eating a physician-supervised diet
* Have other problems that might interfere with ability to participate

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in measures of body weight, body circumferences, and estimated body composition | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Titchenal, PhD, Principal Investigator — Human Nutrition, Food & Animal Sci / Univ of Hawaii; Joannie C Dobbs, PhD, Principal Investigator — Human Nutrition, Food & Animal Sci / Univ of Hawaii
Locations (1):
- Univ of Hawaii Dept of Human Nutrition, Food & Animal Sci, Honolulu, Hawaii, United States